CLINICAL TRIAL: NCT01589796
Title: Effect of Medial vs Traditional Approach to US-guided Transverse Abdominis Plane (TAP) Blocks on Analgesia After Open Inguinal Hernia Repair
Brief Title: Medial Versus Traditional Approach to US-guided TAP Blocks for Open Inguinal Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stamford Anesthesiology Services, PC (Other)
Collaborators: I-Flow (Industry)
Responsible Party: Principal Investigator, Dr. Vlad Frenk, attending anesthesiologist, Stamford Anesthesiology Services, PC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-0308.03
Record Dates: First submitted 2012-04-26; First posted 2012-05-02 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Abdominal Muscles/Ultrasonography; Adult; Ambulatory Surgical Procedures; Anesthetics, Local/Administration & Dosage; Ropivacaine/Administration & Dosage; Ropivacaine/Analogs & Derivatives; Hernia, Inguinal/Surgery; Humans; Nerve Block/Methods; Pain Measurement/Methods; Pain, Postoperative/Prevention & Control; Ultrasonography, Interventional
Keywords: anesthesia; regional anesthetic techniques: transversus abdominis plane block, ilioinguinal nerve block, iliohypogastric nerve block; surgery, inguinal herniorrhaphy; pain, postoperative; surgery, inguinal hernia repair
MeSH Terms: conditions — Hernia; Pain; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- classic TAP (Active Comparator): classic US-guided TAP block in a space between iliac crest and the costal margin in the region of the anterior axillary line
  Interventions: Procedure: TAP block
- Medial TAP (Active Comparator): US-guided TAP block in a space between iliac crest and the costal margin within 1 inch lateral to transversus abdominis muscle origination
  Interventions: Procedure: TAP block

INTERVENTIONS:
Procedure: TAP block — injection of 20ml of Ropivacaine 0.5% in the proper place once it is identified

SUMMARY:
Pain relief after open inguinal hernia repair could be improved by administration of TAP block or ilioinguinal/iliohypogastric nerve block. It is unclear which one works better. The investigators hypothesize that doing TAP block closer to the middle of the abdomen would result in improved pain relief due to simultaneous block of ilioinguinal/iliohypogastric nerves.

DETAILED DESCRIPTION:
This study is a prospective, open, randomized trial. Subjects will be randomized using a computer-generated table of random numbers into 2 groups to receive pre-incisional ipsilateral ultrasound-guided TAP block using classic or medial approach. Group assignments will be sealed in sequentially numbered, opaque envelopes that would be opened by an anesthesiologist performing the block. The research nurse, not involved with patient care after the subject signed written informed consent, will provide postoperative data collection. Study subjects and other anesthesia care providers will also be blinded to group allocation.

All patients will be premedicated with 1-2mg IV midazolam and 50-150 mcg IV fentanyl. In the OR, propofol infusion will be started at 75mcg/kg/hr and titrated for patient comfort. After patient is adequately sedated, ultrasound guided TAP block will be performed in all subjects using a linear 6-15MHz ultrasound probe on a portable ultrasound machine (SonoSite, Bothell, WA). Classic approach group will receive a TAP block as previously described (Hebbard P, 2007). For the medial approach, once the external oblique abdominal, the internal oblique abdominal, and the transversus abdominal muscles were visualized using the ultrasound transducer between the costal margin and the iliac crest at the level of the anterior axillary line (classic approach), the transducer would be moved medially to the point where internal oblique muscle disappears. The injection target area will be within 1 inch lateral to that point.

The place of needle insertion will be prepped with Chlorhexidine gluconate 2% antiseptic solution, and 21G 90-mm StimuQuik needle (Arrow International, Reading, PA) will be used to inject 20ml of Ropivacaine 0.5% in the proper place once it is identified. Each subject will receive local infiltration with 20ml of Lidocaine1% : Bupivacaine 0.25% 1:1 mix prior to the incision by the surgeon as well as 1000 mg of IV acetaminophen and 8 mg IV dexamethasone intraoperatively.

In the postanesthesia care unit (PACU), the patient will be asked to rate their pain at rest upon arrival and at regular intervals on a 0 to 10 numeric rating scale (NRS), where 0 means no pain and 10 is the worst pain imaginable. Hydromorphone 0.5 mg IV will be administered every 5 minutes to maintain an NRS pain score <4 of 10. In cases of postoperative nausea or vomiting, subjects will receive 4mg IV ondansetron, followed by 12.5 mg IV Diphenhydramine if necessary. The Aldrete Recovery Score will be used to transfer the patients from Phase I of recovery, which focuses on providing a transition from a totally anesthetized state to one requiring less intervention. Aldrete Scoring System assesses respiration, oxygen saturation, consciousness, circulation and activity. Each item is scored on a 0 to 2 scale with higher score representing more advanced recovery. Once the score of 9 or higher is reached, the subjects will be transferred to Phase II recovery, which focuses on preparing the patient for dicharge. At discharge, subjects will be instructed to take a combination of oxycodone 5mg and acetaminophen 325mg orally every 4-6 hours for NRS pain score>4 of 10. Postoperative opioid consumption for the 48 hours will be converted to an equivalent dose of oral hydromorphone.

Subjects will be contacted by telephone by a research nurse or one of the investigators not involved in their care, and will be asked about their pain and amount of pain medication they consumed since discharge or since the last phone call respectively. In case of a potential problem, the matter will be referred to a physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 - 75 years of age undergoing open inguinal hernia repair.
* Ability to read and write English

Exclusion Criteria:

* Patients undergoing other concomitant procedure
* Patients with history of diabetes or chronic steroid use
* Patients with chronic or recent (within 1 week prior to procedure) opioid use.
* Patients without the mental capacity to consent for the procedure/study.
* Patients requiring a translator in order to sign the consent for the procedure/study.
* Patients with a history of allergic reactions to local anesthetics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Analgesic consumption after two above mentioned techniques | 48 hours

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Tully Health Center, Stamford, Connecticut
  - Stamford Hospital, Stamford, Connecticut

REFERENCES:
- [Background] Aveline C, Le Hetet H, Le Roux A, Vautier P, Cognet F, Vinet E, Tison C, Bonnet F. Comparison between ultrasound-guided transversus abdominis plane and conventional ilioinguinal/iliohypogastric nerve blocks for day-case open inguinal hernia repair. Br J Anaesth. 2011 Mar;106(3):380-6. doi: 10.1093/bja/aeq363. Epub 2010 Dec 21. PMID 21177284
- [Background] Fredrickson MJ, Paine C, Hamill J. Improved analgesia with the ilioinguinal block compared to the transversus abdominis plane block after pediatric inguinal surgery: a prospective randomized trial. Paediatr Anaesth. 2010 Nov;20(11):1022-7. doi: 10.1111/j.1460-9592.2010.03432.x. PMID 20964768
- [Background] Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007 Aug;35(4):616-7. No abstract available. PMID 18020088
- [Background] Santos Gde C, Braga GM, Queiroz FL, Navarro TP, Gomez RS. Assessment of postoperative pain and hospital discharge after inguinal and iliohypogastric nerve block for inguinal hernia repair under spinal anesthesia: a prospective study. Rev Assoc Med Bras (1992). 2011 Sep-Oct;57(5):545-9. doi: 10.1590/s0104-42302011000500013. English, Portuguese. PMID 22012289
- [Background] Toivonen J, Permi J, Rosenberg PH. Analgesia and discharge following preincisional ilioinguinal and iliohypogastric nerve block combined with general or spinal anaesthesia for inguinal herniorrhaphy. Acta Anaesthesiol Scand. 2004 Apr;48(4):480-5. doi: 10.1111/j.1399-6576.2004.00346.x. PMID 15025612